CLINICAL TRIAL: NCT06891274
Title: Study on the Lung Aerosol Deposition of Ultrasonic Rock Salt Inhalation Therapy
Brief Title: Pulmonary Deposition of Ultrasound Rock Salt Aerosol Inhalation Therapy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jingen Xia (Other)
Responsible Party: Sponsor-Investigator, Jingen Xia, Clinical Professor, China-Japan Friendship Hospital
Organization: China-Japan Friendship Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2024-HX-175
Record Dates: First submitted 2025-03-12; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: COPD; Asthma Bronchiale; Chronic Bronchitis
Keywords: Ultrasound Rock Salt Aerosol Inhalation Therapy; Pulmonary deposition rate; small volume nebulizer
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- USN before SVN (Experimental): The group that received ultrasonic rock salt aerosol inhalation therapy followed by small-volume nebulized inhalation therapy.
  Interventions: Device: USN before SVN
- SVN before USN (Experimental): The group that received small-volume nebulized inhalation therapy followed by ultrasonic rock salt aerosol inhalation therapy.
  Interventions: Device: SVN before USN

INTERVENTIONS:
Device: USN before SVN — The group that received ultrasonic rock salt aerosol inhalation therapy followed by small-volume nebulized inhalation therapy.
  Arms: USN before SVN
Device: SVN before USN — The group that received small-volume nebulized inhalation therapy followed by ultrasonic rock salt aerosol inhalation therapy.
  Other Names: Group B
  Arms: SVN before USN

SUMMARY:
In the in vitro modeling phase, the investigators plan to use a realistic human upper respiratory tract model and an asymmetric ideal bronchial tree model. By combining 3D printing experiments with CFD simulations, the investigators will investigate the respiratory tract deposition rate and distribution of micro - moist particles in ultrasound rock salt aerosol inhalation therapy. This will be compared with a small - volume nebulizer to verify the effectiveness of ultrasound rock salt aerosol inhalation therapy and lay the foundation for further research on the application of this inhalation technique to other drug formulations.

In the clinical phase, the investigators plan to have subjects inhale radioactive aerosols and use PET/CT imaging technology to assess the deposition rate of aerosol particles in the lungs. By quantitatively analyzing the images, the investigators will study their distribution characteristics in real human bodies to verify the accuracy of the in vitro models and the potential for clinical application.

DETAILED DESCRIPTION:
I. Research Background Respiratory diseases, such as asthma, COPD, cystic fibrosis and other chronic respiratory inflammatory diseases, are major global health problems. WHO data shows respiratory diseases are the world's second - leading cause of death, with rising incidence. These diseases, marked by chronic inflammation, airway obstruction and increased airway reactivity, severely affect patients' quality of life. Traditional treatments include inhaled corticosteroids, long - acting bronchodilators and systemic medications. While effective in symptom control and disease progression, they have limitations like systemic side - effects and low drug deposition efficiency from inhalers.

Ultrasonic rock salt aerosol inhalation therapy uses ultrasonic atomization to convert salt solution into tiny aerosol particles, with advantages like high efficiency, micro - moisture, dry aerosol properties, and physiological effects such as enhanced clearance and anti - inflammation.

It has been preliminarily applied in respiratory disease treatment, showing potential in reducing acute exacerbations and improving patients' quality of life. With technological advances and better understanding of aerosol delivery, this therapy has a promising future in respiratory disease management. Future research should focus on confirming its long - term efficacy and safety, exploring personalized applications and evaluating its role in comprehensive treatment strategies.

II. Research Objectives To clarify the process and state of ultrasonic micro - moist rock salt aerosol entering the airway, verify the advantages of the new inhalation device's effective inhalation deposition rate, and provide a new, convenient and effective inhalation technology for drug delivery.

III. Research Overview 3.1 Overall Research Design and Plan This prospective, randomized, crossover study includes two stages: in - vitro modeling and clinical verification.

3.2 Study Population 3.2.1 Inclusion Criteria

* Healthy volunteers.
* Patients with chronic airway diseases needing aerosol inhalation therapy.

3.2.2 Exclusion Criteria

* Age under 18.
* Declining study participation.
* Needing invasive ventilator support.
* Having artificial airways.
* Chronic liver/kidney dysfunction.
* Allergy to radioactive elements.

3.2.3 Withdrawal Criteria

* Patient's consent withdrawal request.
* Investigator's medical judgment for termination.

3.3 Sample Size and Grouping The study will recruit 6 healthy volunteers and 20 patients, randomly divided into Group A (ultrasonic rock salt aerosol inhalation first, then small - volume nebulization) and Group B (small - volume nebulization first, then ultrasonic rock salt aerosol inhalation).

3.4 Research Steps and Related Tests Stage 1: In - vitro Modeling Using real human upper airway and asymmetric ideal bronchial tree models, combining 3D printing and CFD simulation to study aerosol deposition rates and distributions in ultrasonic rock salt aerosol inhalation, compared with small - volume nebulizers.

* Build CFD models for upper airway particle deposition based on CT scans.
* Create CFD models for bronchial tree particle deposition up to the 17th generation.
* Validate deposition characteristics in a whole airway model.

Stage 2: Clinical Verification Using radioactive aerosols and PET/CT imaging to assess lung deposition rates.

* Collect baseline data: demographics, medical history, biochemistry, pulmonary function, etc.
* Aerosol inhalation: patients inhale aerosols in a separate room, with random order. Use 2ml Ga - 68 EDTA for inhalation.
* PET/CT imaging: after inhalation, perform low - dose CT for attenuation correction and lung ventilation PET acquisition.
* Image analysis: use Fiji software and MorphoLibJ plugin to analyze images, calculate deposition rates and concentrations.

3.5 Endpoint Criteria Primary: In - vitro model lung deposition rate, lung drug deposition rate (percentage of deposited drug in lungs relative to total inhaled dose).

Secondary: Peripheral deposition distribution of aerosol particles, residual volume of inhalation device.

IV. Adverse Event Observation

* Radioactive contamination.
* Adverse events related to ultrasonic rock salt aerosol inhalation: dry mouth, nasal burning, pain, etc.
* Nebulization - related adverse events: bronchospasm, coughing, etc.

V. Statistical Analysis 5.1 Sample Size Estimation Based on previous studies, the estimated sample size is 26.

5.2 Data Analysis Analyze data using R Project for Statistical Computing (v 3.5.2). Use Dunnett's test, Bonferroni - corrected post - hoc tests after Kruskal - Wallis ANOVA. Express results as mean ± SD. Use Spearman's correlation for variable relationships. Statistical significance is set at P < 0.05.

VI. Research Ethics The study protocol, consent forms and related materials must be approved by the ethics committee before commencement. Investigators must submit annual reports and inform the committee of any changes. Any changes must be approved before implementation, except those necessary to eliminate immediate risks to participants.

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteers; Patients with chronic airway disease requiring nebulization therapy.

Exclusion Criteria:

Those aged < 18 years; Refusing to participate in the study; Patients requiring invasive ventilator assisted breathing; Patients with artificial airways. Patients with chronic liver and kidney function injury. Allergic to radioactive elements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-03-31 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
In Vitro Model Pulmonary Deposition Rate | Immediately after nebulization
  Aerosol lung deposition rate calculated by in vitro model
Pulmonary Drug Deposition Rate | Immediately after nebulization
  Defined as the percentage of drug deposition in the lungs, relative to the whole inhalation volume

CONTACTS AND LOCATIONS:
Overall Officials: Jingen Xia, M.D, Study Director — China-Japan Friendship Hospital
Locations (1):
- China-Japan Friendship Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang ST, Bao C, Liu Q, Zhang T, Yang Y, Tian X, Zhu Z, Xu KF. Ga-68 EDTA aerosols in evaluation of inhaled-particle deposition and clearance of obstructive pulmonary diseases: A pilot prospective study compared with Galligas. Eur J Clin Invest. 2021 Dec;51(12):e13620. doi: 10.1111/eci.13620. Epub 2021 Jun 2. PMID 34076256
- [Background] Bar-Yoseph R, Kugelman N, Livnat G, Gur M, Hakim F, Nir V, Bentur L. Halotherapy as asthma treatment in children: A randomized, controlled, prospective pilot study. Pediatr Pulmonol. 2017 May;52(5):580-587. doi: 10.1002/ppul.23621. Epub 2016 Oct 10. PMID 27723955
- [Background] Zhang C, Zhu W, Meng Q, Lian N, Wu J, Liu B, Wang H, Wang X, Gu S, Wen J, Shen X, Li Y, Qi X. Halotherapy relieves chronic obstructive pulmonary disease by alleviating NLRP3 inflammasome-mediated pyroptosis. Ann Transl Med. 2022 Dec;10(23):1279. doi: 10.21037/atm-22-5632. PMID 36618788
- [Background] Tanni S, Wehrmeister F, Prudente R, Damatto F, Breda Neto C, Oliveira L, Pagan L, Gatto M, Vieira L, Coelho L, Rezende D, Machado L, Mota G, Gaiato M, Santaella F, Campos E, Franco E, Callegari M, Okoshi MP, Weinreich U. Efficacy of BREATHOX(R) Device Inhalation on Acute Symptoms Associated with COVID-19 (BREATH Study): A Randomized Pilot Clinical Trial. J Clin Med. 2023 Sep 20;12(18):6075. doi: 10.3390/jcm12186075. PMID 37763015